CLINICAL TRIAL: NCT03969004
Title: A Randomized, Placebo-Controlled, Double-Blind Study of Adjuvant Cemiplimab Versus Placebo After Surgery and Radiation Therapy in Patients With High Risk Cutaneous Squamous Cell Carcinoma
Brief Title: Study of Adjuvant Cemiplimab Versus Placebo After Surgery and Radiation Therapy in Patients With High Risk Cutaneous Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R2810-ONC-1788; 2019-000566-38 (EudraCT Number); 2024-511653-22-00 (EU CTIS Number)
Record Dates: First submitted 2019-05-06; First posted 2019-05-31 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cutaneous Squamous Cell Carcinoma
Keywords: High risk
MeSH Terms: interventions — cemiplimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cemiplimab (Experimental)
  Interventions: Drug: Cemiplimab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cemiplimab — Intravenous (IV) infusion over 30 minutes
  Other Names: REGN2810; Libtayo
  Arms: Cemiplimab
Drug: Placebo — Intravenous (IV) infusion over 30 minutes
  Arms: Placebo

SUMMARY:
The primary objective of the study is to compare disease-free survival (DFS) of patients with high-risk cutaneous squamous cell carcinoma (CSCC) treated with adjuvant cemiplimab, versus those treated with placebo, after surgery and radiation therapy (RT).

The secondary objectives of the study are:

* To compare the overall survival (OS) of high-risk CSCC patients treated with adjuvant cemiplimab, versus those treated with placebo, after surgery and RT
* To compare the effect of adjuvant cemiplimab with that of placebo on patients' freedom from locoregional recurrence (FFLRR) after surgery and RT
* To compare the effect of adjuvant cemiplimab with that of placebo on patients' freedom from distant recurrence (FFDR) after surgery and RT
* To compare the effect of adjuvant cemiplimab with that of placebo on the cumulative incidence of second primary CSCC tumors (SPTs) after surgery and RT
* To evaluate the safety of adjuvant cemiplimab and that of placebo in high-risk CSCC patients after surgery and RT
* To assess cemiplimab pharmacokinetics and immunogenicity in human serum

DETAILED DESCRIPTION:
Cemiplimab is a monoclonal antibody. Antibodies are proteins naturally found in the blood. A monoclonal antibody is a special antibody that is manufactured as a medication to target specific proteins in the body that may be involved in cancer. Cemiplimab works by blocking programmed death-1 (PD-1), a cell receptor on immune cells. By blocking PD-1, it is expected that the immune cells will attack cancer cells.

The study is being conducted in participants that have had surgery and radiation therapy for a type of skin cancer called cutaneous squamous cell cancer, and who have a risk that this cancer may come back.

The main purpose of the study is to determine if cemiplimab will prevent cutaneous squamous cell cancer (CSCC) from returning after surgery and radiation. Currently, we know that certain types of CSCC have a high chance of coming back after surgery and radiation. At this time, there is no approved treatment to give patients after surgery and radiation to prevent high-risk CSCC from coming back. We are investigating if the addition of cemiplimab will decrease the chance of these high-risk cancers coming back.

The study will also investigate if cemiplimab may help participants live for longer.

The study has two parts. Part 1: participants will receive every 3 weeks via intravenous infusion (drip into a vein) either cemiplimab (study drug) or placebo (similar to the study drug but without active medicine). After 12 weeks of treatment, cemiplimab or placebo will be given every 6 weeks. Part 1 of the study includes a screening period (up to 28 days), a treatment period (approximately 48 weeks), an end of treatment visit (approximately 30 days after completion of study drug treatment period) and a post-treatment follow-up period (approximately up to 5 years or until skin cancer returns or the study ends).

Part 2 of the study is optional and provides the participant with the option to receive cemiplimab if the cancer comes back if the participant was initially receiving placebo. There is no placebo in Part 2 of the study. If the cancer comes back, the study doctor will discuss with participants if they are eligible to participate in the optional part 2 of the study.

Part 2 of the study includes a brief screening period, a treatment period (approximately 96 weeks) and an end of treatment visit (approximately 30 days after the completion of the study drug treatment period).

ELIGIBILITY:
Key Inclusion Criteria:

* For Japan only, men and women ≥21 years old
* Patient with resection of pathologically confirmed CSCC (primary CSCC lesion only, or primary CSCC with nodal involvement, or CSCC nodal metastasis with known primary CSCC lesion previously treated within the draining lymph node echelon), with macroscopic gross resection of all disease
* High risk CSCC, as defined in the protocol
* Completion of curative intent post-operative radiation therapy (RT) within 2 to 10 weeks of randomization
* Eastern Cooperative Oncology Group performance status (ECOG PS) ≤1
* Adequate hepatic, renal, and bone marrow function as defined in the protocol

Key Exclusion Criteria:

* Squamous cell carcinomas (SCCs) arising in non-cutaneous sites as defined in the protocol
* Concurrent malignancy other than localized CSCC and/or history of malignancy other than localized CSCC within 3 years of date of randomization as defined in the protocol
* Patients with hematologic malignancies (note: patients with chronic lymphocytic leukemia (CLL) are not excluded if they have not required systemic therapy for CLL within 6 months of enrollment)
* Patients with history of distantly metastatic CSCC (visceral or distant nodal), unless the disease-free interval is at least 3 years (regional nodal involvement of disease in draining lymph node basin that was resected and radiated prior to enrollment will not be exclusionary)
* Ongoing or recent (within 5 years of randomization date) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-related adverse events (irAEs). The following are not exclusionary: vitiligo, childhood asthma that has resolved, type 1 diabetes, residual hypothyroidism that required only hormone replacement, or psoriasis that does not require systemic treatment.
* Has had prior systemic anti-cancer immunotherapy for CSCC

Note: Other protocol defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2026-11-03 (Estimated); Study Completion 2028-03-26 (Estimated)

PRIMARY OUTCOMES:
DFS defined as time from randomization to the first documented disease recurrence (local, regional and/or distant); or death due to any cause. | Up to 54 months
  For patients who do not have a tumor recurrence or death, DFS will be censored on the date of last disease assessment.

SECONDARY OUTCOMES:
Overall survival (OS), defined as time from randomization to the date of death. A patient who has not died will be censored on the last known date as alive. | Up to 78 months
FFLRR defined as time from randomization to the date of first locoregional recurrence (LRR). Patients who died without a preceding LRR will be censored on the date of death. | Up to 54 months
  For patients who do not have a LRR or death, FFLRR will be censored on the date of last disease assessment.
Freedom from distant recurrence (FFDR), defined as time from randomization to the date of first distant recurrence (DR). Patients who died without a preceding DR will be censored on the date of death. | Up to 54 months
  For patients who do not have a DR or death, FFDR will be censored on the date of last disease assessment.
Cumulative occurrence of second primary cutaneous squamous cell carcinoma tumor (SPTs) for each patient from randomization to occurrence of first primary endpoint event or end of study. | Up to 54 months
Incidence and severity of treatment-emergent adverse events (TEAE) | Up to 78 months
Incidence of deaths | Up to 78 months
Incidence of laboratory abnormalities | Up to 78 months
Cemiplimab concentrations in serum | Up to 78 months
Anti-drug antibodies (ADA) in serum | Up to 78 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (166):
- United States (40):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Regeneron Study Site, Tucson, Arizona
  - The Angeles Clinic, Los Angeles, California
  - University of Southern California (USC), Los Angeles, California
  - Stanford Cancer Institute, Stanford Medicine at Stanford University, Palo Alto, California
  - University Of California San Francisco (UCSF) - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - George Washington University School of Medicine and Health Sciences, Washington D.C., District of Columbia
  - University of Florida Health, Gainesville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - University of South Florida (USF) - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Regeneron Study Site, Atlanta, Georgia
  - Regeneron Study Site, Chicago, Illinois
  - Regeneron Study Site, Louisville, Kentucky
  - Regeneron Study Site, Baltimore, Maryland
  - Massachusetts General Cancer Center, Boston, Massachusetts
  - Dana Farber/Harvard Cancer Center, Boston, Massachusetts
  - Michigan Medicine- University of Michigan, Ann Arbor, Michigan
  - University of Missouri Health Care - University Physicians - Medicine Specialty Clinic, Columbia, Missouri
  - Washington University in Saint Louis, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Memorial Sloan Kettering, Basking Ridge, New Jersey
  - Memorial Sloan Kettering, Middletown, New Jersey
  - Memorial Sloan Kettering, Montvale, New Jersey
  - Memorial Sloan Kettering, New Brunswick, New Jersey
  - Memorial Sloan Kettering, Commack, New York
  - Memorial Sloan Kettering, Harrison, New York
  - NYU Langone Health, New York, New York
  - Columbia University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering, Uniondale, New York
  - Regeneron Research Site, Cincinnati, Ohio
  - The Ohio State University, Gahanna, Ohio
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology - Baylor Charles A. Simmons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University Of Virginia Health System, Charlottesville, Virginia
- Australia (30):
  - The Border Cancer Hospital Dispensary - Albury Wodonga Regional Cancer Centre, Albury, New South Wales
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - Central Coast Cancer Centre-Gosford and Wyong Hospitals, Gosford, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - North Shore Private Hospital, St Leonards, New South Wales
  - Cancer Care Associates (CCA) Riverina Cancer Care Centre (RCCC), Wagga Wagga, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Illawarra Cancer Care Centre (ICCC), Wollongong, New South Wales
  - Melanoma Institute, Sydney, North South Wales
  - Wide Bay Hospital and Health Service - Cancer Care Services, Bundaberg, Queensland
  - Cairns Hospital, Cairns, Queensland
  - The Royal Brisbane and Women's Hospital, Herston, Queensland
  - ICON Cancer Care, Southport, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Genesis Care Tugun - John Flynn Private Hospital, Tugun, Queensland
  - Wide Bay Hospital and Health Service - Cancer Care Services - Hervey Bay, Urraween, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Ashford Cancer Centre Research-Adelaide Cancer Centre, Kurralta Park, South Australia
  - Royal Hobart Hospital-Hobart Hospital, Hobart, Tasmania
  - Royal Hobart Hospital, Hobart, Tasmania
  - Bendigo Health, Bendigo, Victoria
  - St. Vincent's Hospital, Fitzroy, Victoria
  - Olivia Newton -John Cancer Wellness & Research Centre, Heidelberg, Victoria
  - Peter Maccallum Cancer Centre (PMCC), Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Adelaide Hospital, Adelaide
  - Liverpool Cancer Therapy Center, Liverpool
  - University of New South Wales (UNSW) - Liverpool Hospital - Liverpool Cancer Therapy Centre, Liverpool
  - The Townsville Hospital and Health Service, Townsville
- Belgium (2):
  - Universitair Ziekenhuis Leuven Gasthuisberg Campus, Leuven, Vlaams-Brabant
  - Cliniques Universitaires Saint-Luc, Brussels
- Brazil (11):
  - Fundacao Sao Francisco Xavier - Hospital Marcio Cunha (HMC) - Unidade I, Ipatinga, Minas Gerais
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos, Porte Alegre
  - Instituto Nacional de Cancer Jose Alencar Gomes da Silva ¿ INCA, Santo Cristo, Rio de Janiero
  - Hospital Sao Vicente de Paulo (HSVP), Passo Fundo, Rio Grande do Sul
  - Centro de Pesquisa em Oncologia - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Centro De Novos Tratamentos Itajai, Itajaí, Santa Catarina
  - ANIMI, Lages, Santa Catarina
  - Centro Oncologico Mogi das Cruzes, Mogi das Cruzes, São Paulo
  - Hospital das Clinicas da Faculdade de Medician de Ribeirao Preto FMRP USP, Ribeirão Preto, São Paulo
  - Ynova pesquisa clinica, Florianópolis
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo
- University Health Network- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- France (13):
  - Centre Hospitalier Universitaire (CHU) de Dijon - Hopital du Bocage, Dijon, Dijon Cedex
  - Hopital Saint Andre - CHU de Bordeaux, Bordeaux
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - Centre Hospitalier Universitaire De Grenoble- Hopital Albert Michallon, La Tronche
  - Centre Hospitalier Regional Universitaire de Lille - Hopital Claude Huriez, Lille
  - Centre Leon-Berard (CLB) - Centre de Recherche en Cancerologie Lyon-Est (CRCL), Lyon
  - Centre Hospitalier Universitaire de Nantes (CHU de Nantes) - Hopital Hotel Dieu, Nantes
  - Centre Hospitalier Universitaire de Nice,Hopital l Archet, Nice
  - CIC Cochin Pasteur, Hopital Cochin, Paris
  - Hospital Saint-Louis - APHP, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Rouen-Hopital Charles Nicolle, Rouen
  - Institut Gustave Roussy-Gustave Roussy Cancer Center -DITEP, Villejuif
- Germany (12):
  - NCT Dermatoonkologie -Hautklinik Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitaetsmedizin der Johannes Gutenberg Universitaet Mainz KoeR, Mainz, Rhineland-Palatinate
  - Charite- Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinikum der Ruhr Universitaet Bochum (UKRUB), St. Josef Hospital, Bochum
  - Elbekliniken Buxtehude, Buxtehude
  - Klinikum der Universitaet zu Koeln, Cologne
  - University Hospital Dresden, Dresden
  - Universitaetsklinikum Essen (AoR), Essen
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Universitaetsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - LMU Munchen, München
  - University Hospital Tuebingen, Tübingen
- Greece (2):
  - University of Athens - Hospital of Venereology Dermatology Diseases Andreas Syggros, Athens, Attica
  - Office of Dr. Aimilios Lallas MD, Thessaloniki
- Ireland (3):
  - St. Vincent's University Hospital, Dublin, Leinster
  - University College Cork-Cork University Maternity Hospital, Cork
  - University Hospital Galway, Galway
- Italy (12):
  - ASST Papa Giovanni XXIII, Bergamo
  - Policlinico S.Orsola-Malpighi U.O. Dermatologia - University of Bologna, Bologna
  - ASST Spedali Civili Brescia, Brescia
  - University of Brescia, Brescia
  - Universita di Firenze - Azienda Sanitaria Firenze, Florence
  - University L'Aquila, L’Aquila
  - IRCCS-Istituto Europeo di Oncologia, Milan
  - UOC Oncoematologia AOU Luigi Vanvitelli, Naples
  - U.O.S.C Di Oncologia Medica E Terapie Innovative, Napoli
  - A. Gemelli University Hospital, Catholic University of the Sacred Heart, Rome
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - AOU Citta della Salute e della Scienza di Torino, Torino
- Japan (5):
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Shizuoka Cancer Center - Oncology, Nagaizumi-Cho, Shizuoka
  - National Cancer Center Hospital - Gastrointestinal Oncology, Chuo-ku, Tokyo
  - Niigata Cancer Center Hospital, Niigata
  - Osaka International Cancer Institute - Clinical Oncology, Osaka
- New Zealand (2):
  - Regeneron Study Site, Auckland
  - Palmerston North Hospital, Palmerston North
- Poland (5):
  - Narodowy Instytut Onkologii im. Marii Sk¿odowskiej-Curie - Panstwowy Instytut Badawczy, Oddzial w Gliwicach, Gliwice
  - Regeneron Study Site, Krakow
  - Regeneron Study Site, Poznan
  - Regeneron Study Site, Warsaw
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy, Warsaw
- Russia (7):
  - State Healthcare Institution Oncology Dispensary 2 Ministry of Healthcare of Krasnodar Region, Sochi, Krasnodarskiy Kray
  - SBHI of Stavropol Region Pyatigorsk Interdistrict Oncology Dispensary, Pyatigorsk, Stavropol Kray
  - Regeneron Study Site, Magnitogorsk
  - N.N.Blokhin Cancer Research Center, Moscow
  - Regeneron Research Site, Omsk
  - Federal State Budgetary Institution Rostov Research Institute of Oncology of the Ministry of Healthcare of the Russian Federation, Rostov-on-Don
  - Regeneron Study Site, Saint Petersburg
- Spain (14):
  - Hospital Universitari Vall d'Hebron, Barcelona, Catalonia
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Hospital Universitario de Torrejon, Torrejón de Ardoz, Madrid
  - Catalan institute of Oncology Badalona, Badalona
  - Hospital Clinic de Barcelona - Institut Clinic de Malalties Hematologiques i Oncologiques (ICMHO), Barcelona
  - Genesis Care hospital San Francisco de Asis, Madrid
  - Hospital General Universitario Gregorio Maranon (HGUGM), Madrid
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario 12 de Octubre-Centro de Actividades Ambulatorias, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena-merge, Seville
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Universitario y Politecnico La Fe-merge, Valencia
- United Kingdom (7):
  - Derriford Hospital, Plymouth, Devon
  - University Hospitals Bristol NHS Foundation Trust - Bristol Haematology And Oncology Centre (BHOC) - Bristol Cancer Institute, Bristol, Somerset
  - Velindre NHS Trust, Velindre Cancer Centre, Cardiff
  - The Lothian University Hospitals NHS Lothian - Western General Hospital (WGH), Edinburgh
  - Beatson West of Scotland Cancer Centre - Greater Glasgow Health Board, Glasgow
  - St George's Hospital - St George's University Hospitals NHS Foundation Trust, London
  - The Christie - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- [Derived] Rischin D, Porceddu S, Day F, Brungs DP, Christie H, Jackson JE, Stein BN, Su YB, Ladwa R, Adams G, Bowyer SE, Otty Z, Yamazaki N, Bossi P, Challapalli A, Hauschild A, Lim AM, Patel VA, Walker JL, De Liz Vassen Schurmann M, Queirolo P, Canueto J, Ferreira da Silva FA, Stratigos A, Guminski A, Lin C, Damian F, Flatz L, Taylor AE, Carr DR, Harris S, Kirtbaya D, Quereux G, Rutkowski P, Basset-Seguin N, Khushalani NI, Robert C, Ju H, Joseph C, Bansal S, Chen CI, Seebach F, Yoo SY, Lowy I, Goncalves P, Fury MG; C-POST Trial Investigators. Adjuvant Cemiplimab or Placebo in High-Risk Cutaneous Squamous-Cell Carcinoma. N Engl J Med. 2025 Aug 21;393(8):774-785. doi: 10.1056/NEJMoa2502449. Epub 2025 May 31. PMID 40454639
- See also: Related Info — https://c-poststudy.com/